CLINICAL TRIAL: NCT07016061
Title: Acute Effects of Motor Imagery and Action Observation in the Elderly: Single-Blind Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, tolunay keskin, PhD Student, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/16-20
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Elderly (People Aged 65 or More)
Keywords: imagery; Mirror Neurons; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be divided into five groups: a motor imagery group, an action observation group, an exercise group, a combined exercise group, and a control group.
Who Masked: Outcomes Assessor
Masking Description: The study will be conducted as a single-blind randomized controlled trial. Participants will be randomly assigned to one of five groups, and outcome assessments will be performed by an evaluator who is blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Motor İmagery Group (Active Comparator): Motor imagery is the mental simulation of movement without actual physical execution. Participants will engage in a motor imagery exercise program consisting of 5 minutes of warm-up, 20 minutes of motor imagery, and 5 minutes of cool-down, totaling 30 minutes.
  Interventions: Other: Motor İmagery Group
- Action Observation Group (Active Comparator): Participants will receive an action observation training program delivered by researchers, including 5 minutes of warm-up, 20 minutes of action observation, and 5 minutes of cool-down, totaling 30 minutes.
  Interventions: Other: Action Observation Group
- Exercise Group (Active Comparator): Participants will perform a standard physical exercise program. The session will last 30 minutes, including warm-up, exercise, and cool-down phases.
  Interventions: Other: Exercise Group
- Combined Group (Motor Imagery + Action Observation+Exercise) (Active Comparator): Participants will engage in a combined motor imagery and action observation program for a total of 30 minutes, incorporating elements of both interventions.
  Interventions: Other: Combined Group (Motor Imagery + Action Observation+Exercise)
- Control Group (No Intervention): Participants will not receive any intervention during the study period. After the completion of the 3-session evaluation phase, they will be given the option to participate in the exercise program if they wish.

INTERVENTIONS:
Other: Motor İmagery Group — Participants will engage in a motor imagery exercise program consisting of 5 minutes of warm-up, 20 minutes of motor imagery, and 5 minutes of cool-down, totaling 30 minutes. The intervention will be administered in three sessions per week for one week.
  Arms: Motor İmagery Group
Other: Action Observation Group — Participants will receive an action observation training program delivered by researchers, including 5 minutes of warm-up, 20 minutes of action observation, and 5 minutes of cool-down, totaling 30 minutes. The intervention will be administered in three sessions per week for one week.
  Arms: Action Observation Group
Other: Exercise Group — Participants will perform a standard physical exercise program. The session will last 30 minutes, including warm-up, exercise, and cool-down phases. The intervention will be administered in three sessions per week for one week.
  Arms: Exercise Group
Other: Combined Group (Motor Imagery + Action Observation+Exercise) — articipants will engage in a combined motor imagery and action observation program for a total of 30 minutes, incorporating elements of both interventions. The intervention will be administered in three sessions per week for one week.
  Arms: Combined Group (Motor Imagery + Action Observation+Exercise)

SUMMARY:
The aim of this study is to investigate the effects of acute action observation, motor imagery, exercise, and combined exercise training on parameters such as balance, reaction time, flexibility, fear of falling, cognitive status, attention, and memory in older adults.

DETAILED DESCRIPTION:
Previous studies investigating motor imagery and action observation training have examined their long-term effects in both young and older adults. Existing evidence regarding the benefits of exercise training indicates positive effects in both populations. However, the number of studies focusing on the acute effects of motor imagery and action observation training in the literature is very limited. Individuals who meet the inclusion criteria will be randomly assigned-using the Research Randomizer application-into five groups: motor imagery, action observation, exercise, combined exercise, and control group. A total of 50 participants, with 10 individuals in each group, will be included in the study. Assessments will be conducted before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 65 years or older, Female gender, Literate in Turkish, Scoring 21 or above on the Montreal Cognitive Assessment (MoCA) Version 7.1, No health conditions that would prevent participation in exercise

Exclusion Criteria:

* Presence of serious health problems that would prevent participation in the study (e.g., trauma, cancer, surgery, severe cardiac or musculoskeletal disorders)

Participation in other intervention trials or observational studies during the intervention period, or initiation of a physical exercise program within 2 weeks following the intervention period

Any medical condition or chronic medication use that may jeopardize safety or affect cognitive functions (e.g., neuroleptics)

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Female
Enrollment: 50 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test | 2 weeks
  The Timed Up and Go (TUG) test is a simple and widely used clinical test to assess functional mobility, balance, and fall risk in older adults. It measures the time it takes for an individual to stand up from a chair, walk three meters, turn around, walk back, and sit down.

SECONDARY OUTCOMES:
Functional Reach Test (FRT) | 2 weeks
  The Functional Reach Test (FRT) is a clinical assessment tool used to evaluate dynamic balance and stability. It measures the maximum distance an individual can reach forward beyond arm's length while standing in a fixed position without losing balance or taking a step.
10-Meter Walk Test (10MWT) | 2 weeks
  The 10-Meter Walk Test (10MWT) is a standardized assessment used to measure walking speed over a short distance. It evaluates functional mobility, gait performance, and lower extremity motor function by recording the time taken to walk a distance of 10 meters at a comfortable or maximum pace.
Computerized Serial Reaction Time Test (SRTT) | 2 weeks
  The Computerized Serial Reaction Time Test (SRTT) is a cognitive-motor task used to assess implicit motor learning, reaction time, and attention. In this test, participants respond as quickly and accurately as possible to visual stimuli that appear in a specific sequence on a computer screen, allowing for the measurement of both response speed and learning patterns
Five Times Sit-to-Stand Test (FTSST) | 2 weeks
  The Five Times Sit-to-Stand Test (FTSST) is a simple and reliable clinical assessment used to evaluate lower limb muscle strength, functional mobility, and fall risk. It measures the time it takes for an individual to rise from a chair and sit back down five times as quickly as possible without using their arms for support
Back Scratch Test | 2 weeks
  The Back Scratch Test is a flexibility assessment used to measure the range of motion and flexibility of the upper body, particularly the shoulders. It involves reaching one hand over the shoulder and the other behind the back to see how close the fingers can come to each other, or whether they overlap.
Falls Efficacy Scale International, FES-I | 2 weeks
  The Falls Efficacy Scale-International (FES-I) is a validated questionnaire designed to assess fear of falling in older adults. It measures the level of concern individuals have about falling during a range of daily activities, both inside and outside the home. Higher scores indicate greater fear of falling.
Montreal Cognitive Assessment (MoCA) | 2 weeks
  The Montreal Cognitive Assessment (MoCA) is a widely used screening tool designed to detect mild cognitive impairment. It assesses various cognitive domains including attention, executive functions, memory, language, visuospatial skills, and orientation. The test provides a total score out of 30, with higher scores indicating better cognitive performance.
Trail Making Test | 2 weeks
  The Trail Making Test (TMT) is a neuropsychological assessment used to evaluate visual attention, processing speed, and executive function. It consists of two parts: Part A requires connecting numbered dots in sequence, while Part B involves alternating between numbers and letters in order. The time taken to complete each part is recorded, with longer times indicating potential cognitive impairment
Verbal Memory Processes Test | 2 weeks
  The Verbal Memory Processes Test is a neuropsychological assessment designed to evaluate various aspects of verbal memory, including encoding, storage, and retrieval of verbal information. It typically involves tasks such as recalling word lists, story recall, or recognizing verbal stimuli to assess immediate and delayed memory performance

CONTACTS AND LOCATIONS:
Overall Officials: tolunay keskın, Phd Student, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylül University, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not consent to the use of my data